CLINICAL TRIAL: NCT00927680
Title: Familial Colorectal Cancer In Puerto Rico: A Feasibility Study
Brief Title: Familial Colorectal Cancer Registry in Hispanics
Acronym: PURIFICAR
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Puerto Rico (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Marcia R. Cruz-Correa, MD, PhD, Associate Professor of Medicine, Biochemistry and Surgery at University of Puerto Rico School of Medicine, Director of Gastrointestinal Oncology at the University of Puerto Rico (UPR) Comprehensive Cancer Center, University of Puerto Rico
Other Study IDs: R03CA130034 NCI; R03CA130034 (NIH)
Record Dates: First submitted 2009-06-24; First posted 2009-06-25 (Estimated); Last update posted 2020-11-19 (Actual); Status verified 2020-11

CONDITIONS: Colorectal Cancer; Gastric Cancer; Colorectal Neoplasms; Colorectal Adenoma; Lynch Syndrome
Keywords: Colorectal Cancer; Familial Colorectal Cancer; Genetics; Hispanics; Lynch Syndrome
MeSH Terms: conditions — Colorectal Neoplasms; Stomach Neoplasms; Colorectal Neoplasms, Hereditary Nonpolyposis

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Tumor blocks (colorectal tumors) and blood samples
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Colorectal cancer cases
- Controls

SUMMARY:
Colorectal cancer (CRC) is the second leading cause of cancer in Puerto Rico (PR) accounting for approximately 1,500 individuals annually, which represent 12% of all cancer cases in the island. The genetic epidemiology of CRC among Hispanic populations is not well studied, hence studies focused on large, well defined ethnic groups such as Puerto Ricans, are clearly warranted. The first step towards evaluating the molecular, environmental, and genetic epidemiology of CRC in PR is to establish a population-based familial CRC registry. The following specific aims have been proposed:

Specific Aim 1: To prospectively identify and recruit approximately 300 CRC probands from two distinct geographical areas in PR (Metropolitan and Southern Region). From each proband the investigators will obtain a pedigree extended to second-degree relatives and cousins. Assuming 10% will be positive for a family history of CRC, the investigators will then recruit all 30 probands with a family history of CRC and a sample of 15 family-history negative probands and obtain: paraffin-embedded tumors blocks, blood samples, risk factor and food frequency questionnaires.

Specific Aim 2: To prospectively identify and recruit selected relatives (parents, grandparents, and same generation relatives - cousins and siblings) from the 45 probands identified in Specific Aim 1. In addition, for siblings and cousins of probands (i.e. relatives in the same generation as the proband), the investigators will obtain risk factor and food frequency questionnaires, and for colorectal cancer cases, tumor blocks and pathology reports of their cancers.

Specific Aim 3: To estimate from this pilot study the following parameters: (a) response rate of probands and their selected relatives; (b) response rate of participants for each data item; (c) family history of CRC and other cancers; (d) number of living first- and second-degree relatives and cousins of probands; (e) number of these relatives who live in the same household and region/municipality; (f) prevalence/distribution of selected risk factors from the administered questionnaires.

DETAILED DESCRIPTION:
Data obtained from this study will serve as the foundation for our large, island-wide, population-based, genetic-epidemiologic study of familial colorectal cancer in Puerto Rico. Through this feasibility study, we will assess the feasibility: (1) of recruiting colorectal cancer patients using the PR Central Cancer Registry, (2) of evaluating family pedigrees and recruiting the relatives of probands (3) obtaining tumor, blood, medical and exposure information from both probands and their relatives. Providing important data on Hispanic populations that would enable family-based case-control studies of risk factors for CRC, with an emphasis on candidate genes in selected carcinogenic pathways, genetic and epigenetic modifications. Furthermore, information obtained from this proposal may serve to identify families that would be informative for linkage studies to potentially map new genes, evaluate genotype-phenotype correlations, gene-gene and gene-environmental interactions.

ELIGIBILITY:
Inclusion criteria:

* patients with colon polyps or colon cancer
* patients will have a colonoscopy or colon surgery to treat a benign condition such as fissure, fistula, or hemorrhoids

Exclusion criteria:

Participation in this study is limited to persons 15 years or older with colon polyps or colon cancer and control subjects 21 years or older with no malignant conditions in the colon and / or rectum. Controls between the ages of 15 to 20 years will be not evaluated. The reason is colon cancer occurs in people under 21 years, except in special cases associated with certain genetic causes. People who cannot sign the consent may not participate in this study.

Min Age: 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: 1. Probands will be ascertained from the Puerto Rico Central Cancer Registry (PRCCR), from the monthly report of incident colorectal cancer cases. Eligible cases were persons (1) with pathologic diagnosis of colorectal cancer; (2) who were 15 years of age or older, and (3) without previous history of colorectal cancer.
  2. Probands will be ascertained from the Oncology Hospital, UDH Hospital and the Ashford Presbyterian Community Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2007-07; Primary Completion 2025-12 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
We will recruit individuals with colorectal cancer with and without family history of CRC and their immediate family members and obtain the following: paraffin-embedded tumors blocks, blood samples, risk factor and food frequency questionnaires. | 10 years

SECONDARY OUTCOMES:
We will study the following parameters that we help us plan the larger population-based study such as: response rate of probands and their selected relatives, response rate of participants (probands and relatives), etcetera. | 10 years

CONTACTS AND LOCATIONS:
Overall Officials: Marcia R. Cruz-Correa, MD, PhD, Principal Investigator — University of Puerto Rico
Locations (2):
- Puerto Rico (2):
  - Oncologic Hospital, San Juan, PR
  - University of Puerto Rico Comprehensive Cancer Center, San Juan